CLINICAL TRIAL: NCT00838565
Title: Phase 1, Randomized, Patient And Investigator-blind, Placebo-controlled Study To Investigate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Multiple Intravenously Administered Doses Of Pf-04236921 In Patients With Rheumatoid Arthritis Receiving Methotrexate
Brief Title: Phase I Study Of The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Multiple Intravenously Administered Doses Of PF-04236921 In Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: B0151002; 2009-009866-15 (EudraCT Number)
Record Dates: First submitted 2009-02-04; First posted 2009-02-06 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Safety and tolerability Pharmacokinetics Pharmacodynamics PF-04236921
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PF-04236921 (Experimental)
  Interventions: Drug: dose level 1; Drug: dose level 2; Drug: dose level 3; Drug: dose level 4

INTERVENTIONS:
Drug: Placebo — intravenous infusion on three consecutive months
  Arms: Placebo
Drug: dose level 1 — intravenous infusion on three consecutive months
  Arms: PF-04236921
Drug: dose level 2 — intravenous infusion on three consecutive months
  Arms: PF-04236921
Drug: dose level 3 — intravenous infusion on three consecutive months
  Arms: PF-04236921
Drug: dose level 4 — intravenous infusion on 3 consecutive months
  Arms: PF-04236921

SUMMARY:
This study will evaluate the safety and tolerability of PF-04236921 administered monthly as three intravenous infusions. Each group of patients will be assigned to a dose level; Safety and tolerability of a low dose level will be required before proceeding to successively higher dose levels. Blood tests will be performed to measure the amount of drug and changes in measures of inflammation.

DETAILED DESCRIPTION:
Safety and Tolerability and Pharmacokinetic/Pharmacodynamic assessment of inflammation-related biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid Arthritis on a stable dose of methotrexate
* Rheumatoid Arthritis disease activity as assessed by blood tests

Exclusion Criteria:

* Serious or uncontrolled medical conditions
* Current or recent treatment with disease-modifying drugs other than methotrexate including but not limited to leflunomide, sulfasalazine, etanercept, infliximab, adalimumab, abatacept, rituximab
* Current oral glucocorticoid dose of more than 10 mg/d prednisone equivalent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-05-20 (Actual); Primary Completion 2012-02-02 (Actual); Study Completion 2012-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (3):
  - Allergy, Asthma, Arthritis, & Lung, Daytona Beach, Florida
  - Millennium Research, Ormond Beach, Florida
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
- South Korea (3):
  - Inha University Hospital, Medicine/Rheumatology, Incheon
  - Seoul National University Hospital, Rheumatology, Internal Medicine, Seoul
  - Yonsei University College of Medicine, Severance Hospital, Clinical Trial Center, Seoul
- Spain (2):
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, A Coruña
  - Complexo Hospitalario Universitario A Coruña, A Coruña

REFERENCES:
- [Derived] Li C, Shoji S, Beebe J. Pharmacokinetics and C-reactive protein modelling of anti-interleukin-6 antibody (PF-04236921) in healthy volunteers and patients with autoimmune disease. Br J Clin Pharmacol. 2018 Sep;84(9):2059-2074. doi: 10.1111/bcp.13641. Epub 2018 Jun 25. PMID 29776017
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0151002&StudyName=Phase%20I%20Study%20Of%20The%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%20And%20Pharmacodynamics%20Of%20Multiple%20Intravenously%20Administered%20Doses%20Of%20PF-042369

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matched to PF-04236921 intravenous infusion over approximately 1 hour on Day 1, 28 and 56. Methotrexate orally or parenterally starting from at least 16 weeks prior to randomization as per local standard-of-care practice followed by a stable dose of methotrexate between 7.5 to 25 mg per week from at least 6 weeks prior to randomization to Day 84. Participants were followed up to 624 days.
- PF-04236921 1 mg: PF-04236921 1 mg intravenous infusion over approximately 1 hour on Day 1, 28 and 56. Methotrexate orally or parenterally starting from at least 16 weeks prior to randomization as per local standard-of-care practice followed by a stable dose of methotrexate between 7.5 to 25 mg per week from at least 6 weeks prior to randomization to Day 84. Participants were followed up to 624 days.
- PF-04236921 10 mg: PF-04236921 10 mg intravenous infusion over approximately 1 hour on Day 1, 28 and 56. Methotrexate orally or parenterally starting from at least 16 weeks prior to randomization as per local standard-of-care practice followed by a stable dose of methotrexate between 7.5 to 25 mg per week from at least 6 weeks prior to randomization to Day 84. Participants were followed up to 624 days.
- PF-04236921 30 mg: PF-04236921 30 mg intravenous infusion over approximately 1 hour on Day 1, 28 and 56. Methotrexate orally or parenterally starting from at least 16 weeks prior to randomization as per local standard-of-care practice followed by a stable dose of methotrexate between 7.5 to 25 mg per week from at least 6 weeks prior to randomization to Day 84. Participants were followed up to 624 days.
- PF-04236921 100 mg: PF-04236921 100 mg intravenous infusion over approximately 1 hour on Day 1, 28 and 56. Methotrexate orally or parenterally starting from at least 16 weeks prior to randomization as per local standard-of-care practice followed by a stable dose of methotrexate between 7.5 to 25 mg per week from at least 6 weeks prior to randomization to Day 84. Participants were followed up to 624 days.
- PF-04236921 250 mg: PF-04236921 250 mg intravenous infusion over approximately 1 hour on Day 1, 28 and 56. Methotrexate orally or parenterally starting from at least 16 weeks prior to randomization as per local standard-of-care practice followed by a stable dose of methotrexate between 7.5 to 25 mg per week from at least 6 weeks prior to randomization to Day 84. Participants were followed up to 624 days.
Period: Overall Study
Arm/Group | Placebo | PF-04236921 1 mg | PF-04236921 10 mg | PF-04236921 30 mg | PF-04236921 100 mg | PF-04236921 250 mg
Started | 9 | 7 | 6 | 6 | 6 | 7
Treated | 9 | 6 | 6 | 6 | 6 | 7
Completed | 9 | 4 | 5 | 6 | 6 | 5
Not Completed | 0 | 3 | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 2
Not completed — Other | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Randomized but not Treated | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-04236921 1 mg | PF-04236921 10 mg | PF-04236921 30 mg | PF-04236921 100 mg | PF-04236921 250 mg | Total
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 6 | 7 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (8.5) | 61.7 (7.9) | 49.8 (13.5) | 46.0 (4.1) | 56.7 (8.9) | 55.4 (9.8) | 55.2 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 5 | 5 | 4 | 6 | 34
  Male | 1 | 0 | 1 | 1 | 2 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study medication and up to 28 days after last dose or until serum PF-04236921 concentrations were below the LLOQ that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline up to 28 days after last dose of study medication or until serum PF-04236921 concentrations below the LLOQ (up to Day 624)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04236921 1 mg | PF-04236921 10 mg | PF-04236921 30 mg | PF-04236921 100 mg | PF-04236921 250 mg
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 6 | 7
participants
  AEs | 9 | 4 | 4 | 6 | 6 | 5
  SAEs | 0 | 0 | 0 | 2 | 1 | 0

2. Primary Outcome: Number of Participants With Positive Anti-drug Antibodies Response
Time Frame: Day 1, 28, 56, 84, 174, 354, End of Study (Day 624)
Population: Safety analysis set included all participants who received at least 1 dose of study medication. Here 'n' signifies those participants who were evaluable for this measure at specified time points for each arm, respectively.
Measure: Number; unit: participants
Arm/Group | PF-04236921 1 mg | PF-04236921 10 mg | PF-04236921 30 mg | PF-04236921 100 mg | PF-04236921 250 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7
participants
  Day 1 | 0 | 0 | 0 | 0 | 0
  Day 28: number analyzed (Participants) | 6 | 5 | 6 | 6 | 7
  Day 28 | 0 | 0 | 0 | 0 | 0
  Day 56: number analyzed (Participants) | 6 | 5 | 6 | 6 | 7
  Day 56 | 0 | 0 | 0 | 0 | 0
  Day 84: number analyzed (Participants) | 6 | 5 | 6 | 6 | 7
  Day 84 | 0 | 0 | 0 | 0 | 0
  Day 174: number analyzed (Participants) | 2 | 5 | 4 | 6 | 7
  Day 174 | 0 | 0 | 0 | 0 | 0
  Day 354: number analyzed (Participants) | 0 | 1 | 5 | 6 | 5
  Day 354 |  | 0 | 0 | 0 | 0
  End of Study: number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
  End of Study | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Maximum Observed Serum Concentration (Cmax): Day 1
Time Frame: Day 1: Pre-dose (0 hour), 15 minutes, 168 hours, 336 hours post-dose
Population: Pharmacokinetic (PK) parameter analysis population included all enrolled and treated participants who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-04236921 1 mg | PF-04236921 10 mg | PF-04236921 30 mg | PF-04236921 100 mg | PF-04236921 250 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7
nanogram per milliliter (ng/mL) | 421.6 (162.89) | 4631 (1429.9) | 11320 (2167.2) | 42290 (7883.0) | 66280 (59405)

4. Primary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax): Day 1
Time Frame: Day 1: Pre-dose (0 hour), 15 minutes, 168 hours, 336 hours post-dose
Population: PK parameter analysis population included all enrolled and treated participants who had at least 1 of the PK parameters of interest.
Measure: Median (Full Range); unit: days
Arm/Group | PF-04236921 1 mg | PF-04236921 10 mg | PF-04236921 30 mg | PF-04236921 100 mg | PF-04236921 250 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7
days | 0.0521 [0.0521 to 0.0528] | 0.0521 [0.0521 to 0.0521] | 0.0521 [0.0521 to 0.0521] | 0.0521 [0.0278 to 0.0521] | 0.0521 [0.0521 to 0.0528]

5. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-168)]: Day 1
Description: AUC (0-168) = Area under the serum concentration versus time curve from time zero (pre-dose) to 168 hours (0-168).
Time Frame: Day 1: Pre-dose (0 hour), 15 minutes, 168 hours post-dose
Population: as for outcome 4
Measure: Geometric Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | PF-04236921 1 mg | PF-04236921 10 mg | PF-04236921 30 mg | PF-04236921 100 mg | PF-04236921 250 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7
ng*day/mL | 1899 (1090.1) | 19570 (5335.7) | 54140 (9345.0) | 206000 (40578) | 348500 (336540)

6. Primary Outcome: Maximum Observed Serum Concentration (Cmax): Day 28
Time Frame: Day 28: Pre-dose (0 hour), 15 minutes, 168 hours, 336 hours post-dose
Population: PK parameter analysis population included all enrolled and treated participants who had at least 1 of the PK parameters of interest. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04236921 1 mg | PF-04236921 10 mg | PF-04236921 30 mg | PF-04236921 100 mg | PF-04236921 250 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 7
ng/mL | 617.6 (430.18) | 4719 (1807.2) | 13680 (3453.2) | 57280 (6396.4) | 158300 (50966)

7. Primary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax): Day 28
Time Frame: Day 28: Pre-dose (0 hour), 15 minutes, 168 hours, 336 hours post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: days
Arm/Group | PF-04236921 1 mg | PF-04236921 10 mg | PF-04236921 30 mg | PF-04236921 100 mg | PF-04236921 250 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 7
days | 0.0521 [0.0521 to 0.0528] | 0.0521 [0.0521 to 0.0521] | 0.0521 [0.0521 to 0.0521] | 0.0521 [0.0521 to 0.0528] | 0.0521 [0.0514 to 0.0521]

8. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-168)]: Day 28
Description: AUC (0-168) = Area under the serum concentration versus time curve from time zero (pre-dose) to 168 hours (0-168).
Time Frame: Day 28: Pre-dose (0 hour), 15 minutes, 168 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | PF-04236921 1 mg | PF-04236921 10 mg | PF-04236921 30 mg | PF-04236921 100 mg | PF-04236921 250 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 7
ng*day/mL | 3104 (2369.7) | 21660 (7232.7) | 76510 (19496) | 316900 (45597) | 767900 (213320)

9. Primary Outcome: Maximum Observed Serum Concentration (Cmax): Day 56
Time Frame: Day 56: Pre-dose (0 hour), 15 minutes, 168 hours, 336 hours, 672 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04236921 1 mg | PF-04236921 10 mg | PF-04236921 30 mg | PF-04236921 100 mg | PF-04236921 250 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 7
ng/mL | 741.0 (977.35) | 4424 (1384.8) | 19650 (1537.5) | 64850 (13289) | 164600 (35644)

10. Primary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax): Day 56
Time Frame: Day 56: Pre-dose (0 hour), 15 minutes, 168 hours, 336 hours, 672 hours post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: days
Arm/Group | PF-04236921 1 mg | PF-04236921 10 mg | PF-04236921 30 mg | PF-04236921 100 mg | PF-04236921 250 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 7
days | 0.0521 [0.0521 to 0.0542] | 0.0521 [0.0521 to 0.0521] | 0.0521 [0.0521 to 0.0521] | 0.0521 [0.0521 to 0.0521] | 0.0521 [0.0521 to 0.0528]

11. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-168)]: Day 56
Description: AUC (0-168) = Area under the serum concentration versus time curve from time zero (pre-dose) to 168 hours (0-168).
Time Frame: Day 56: Pre-dose (0 hour), 15 minutes, 168 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | PF-04236921 1 mg | PF-04236921 10 mg | PF-04236921 30 mg | PF-04236921 100 mg | PF-04236921 250 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 7
ng*day/mL | 3730 (4479.8) | 23200 (7558.6) | 101100 (6438.2) | 389100 (71949) | 912200 (209610)

12. Primary Outcome: Serum Decay Half-Life (t1/2): Day 56
Description: Serum decay half-life is the time measured for the serum concentration to decrease by one half.
Time Frame: Day 56: Pre-dose (0 hour), 15 minutes, 168 hours, 336 hours, 672 hours post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: days
Arm/Group | PF-04236921 1 mg | PF-04236921 10 mg | PF-04236921 30 mg | PF-04236921 100 mg | PF-04236921 250 mg
Number analyzed (Participants) | 2 | 5 | 5 | 6 | 6
days | 45.50 (NA) [45.0 to 46.0] | 36.90 (11.010) [19.3 to 49.5] | 45.30 (9.5166) [32.9 to 54.3] | 38.80 (6.9500) [35.5 to 51.7] | 51.70 (9.2230) [31.9 to 59.2]

13. Other Pre Specified Outcome: Change From Baseline in C-Reactive Protein (CRP) Concentrations at Day 7, 14, 28, 35, 42, 56, 63, 70, 84, 129, 174, 219, 264, 309, 354, 399, 444, 489, 534, 579, 624 and Early Discontinuation
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultra sensitive assay. A decrease in the level of CRP indicates reduction in inflammation.
Time Frame: Baseline, Day 7, 14, 28, 35, 42, 56, 63, 70, 84, 129, 174, 219, 264, 309, 354, 399, 444, 489, 534, 579, 624, Early Discontinuation
Population: Pharmacodynamic analysis set included all enrolled participants who received at least 1 dose of study medication and had at least 1 pharmacodynamic parameter. Data collected at Early Discontinuation included those subjects who left the study early.'N' (number of participants analyzed) = participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | Placebo | PF-04236921 1 mg | PF-04236921 10 mg | PF-04236921 30 mg | PF-04236921 100 mg | PF-04236921 250 mg
Number analyzed (Participants) | 9 | 6 | 6 | 5 | 6 | 7
milligram per liter (mg/L)
  Baseline | 11.54 (12.452) | 9.95 (7.886) | 11.01 (6.419) | 7.23 (8.316) | 8.88 (5.797) | 17.91 (25.572)
  Change at Day 7 | -0.09 (7.128) | -6.36 (8.322) | -9.85 (5.830) | -6.43 (7.766) | -8.26 (5.747) | -17.31 (25.317)
  Change at Day 14 | -2.63 (10.877) | -5.81 (9.019) | -10.03 (6.134) | -6.69 (8.357) | -8.56 (5.827) | -17.52 (25.571)
  Change at Day 28: number analyzed (Participants) | 9 | 6 | 5 | 5 | 6 | 7
  Change at Day 28 | 1.06 (5.153) | -4.48 (8.635) | -9.98 (6.168) | -6.70 (8.402) | -8.59 (5.797) | -17.52 (25.634)
  Change at Day 35: number analyzed (Participants) | 9 | 6 | 5 | 5 | 6 | 7
  Change at Day 35 | 0.74 (6.859) | -6.51 (8.817) | -11.10 (6.617) | -6.52 (8.515) | -8.63 (5.824) | -17.56 (25.608)
  Change at Day 42: number analyzed (Participants) | 9 | 6 | 5 | 5 | 6 | 7
  Change at Day 42 | -0.06 (6.823) | -6.60 (8.299) | -11.02 (6.653) | -6.82 (8.384) | -8.65 (5.833) | -17.59 (25.614)
  Change at Day 56: number analyzed (Participants) | 9 | 6 | 5 | 5 | 6 | 7
  Change at Day 56 | -0.07 (6.724) | -6.14 (8.918) | -10.68 (6.503) | -6.65 (8.453) | -8.66 (5.817) | -17.59 (25.611)
  Change at Day 63: number analyzed (Participants) | 9 | 6 | 5 | 5 | 6 | 7
  Change at Day 63 | -0.10 (8.214) | -7.83 (8.284) | -11.35 (6.758) | -6.67 (8.472) | -8.68 (5.812) | -17.58 (25.611)
  Change at Day 70: number analyzed (Participants) | 9 | 6 | 5 | 5 | 6 | 7
  Change at Day 70 | 1.68 (13.334) | -7.67 (8.263) | -11.25 (6.740) | -6.82 (8.441) | -8.69 (5.810) | -17.60 (25.608)
  Change at Day 84: number analyzed (Participants) | 9 | 6 | 5 | 5 | 6 | 7
  Change at Day 84 | 5.16 (26.869) | -6.23 (9.130) | -10.88 (6.555) | -6.88 (8.441) | -8.54 (5.760) | -17.58 (25.587)
  Change at Day 129: number analyzed (Participants) | 8 | 4 | 5 | 5 | 6 | 7
  Change at Day 129 | 5.10 (23.998) | -8.49 (10.327) | -10.26 (5.772) | -6.63 (8.513) | -8.65 (5.840) | -17.66 (25.605)
  Change at Day 174: number analyzed (Participants) | 7 | 2 | 5 | 5 | 6 | 7
  Change at Day 174 | 2.42 (15.773) | -4.55 (0.735) | -8.73 (4.550) | -4.28 (4.545) | -8.57 (5.781) | -17.62 (25.581)
  Change at Day 219: number analyzed (Participants) | 7 | 2 | 5 | 5 | 6 | 6
  Change at Day 219 | 4.35 (18.530) | 4.01 (10.083) | -6.22 (4.790) | -6.40 (8.602) | -8.66 (5.807) | -19.43 (26.221)
  Change at Day 264: number analyzed (Participants) | 6 | 1 | 3 | 4 | 6 | 5
  Change at Day 264 | -5.33 (6.033) | -6.30 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | -4.06 (1.961) | -2.58 (1.056) | -8.07 (5.922) | -16.60 (28.318)
  Change at Day 309: number analyzed (Participants) | 3 | 0 | 2 | 5 | 6 | 5
  Change at Day 309 | -6.19 (7.987) |  | -4.36 (1.761) | -5.80 (8.951) | -7.63 (6.599) | -16.52 (28.364)
  Change at Day 354: number analyzed (Participants) | 3 | 0 | 1 | 5 | 6 | 5
  Change at Day 354 | -3.33 (12.217) |  | -2.30 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | -5.11 (9.482) | -8.12 (5.849) | -16.61 (28.313)
  Change at Day 399: number analyzed (Participants) | 3 | 0 | 0 | 3 | 6 | 5
  Change at Day 399 | -2.49 (8.119) |  |  | -6.47 (8.596) | 4.68 (32.401) | -16.56 (28.330)
  Change at Day 444: number analyzed (Participants) | 1 | 0 | 0 | 1 | 3 | 5
  Change at Day 444 | -15.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. |  |  | -0.79 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | -4.78 (4.694) | -15.57 (28.927)
  Change at Day 489: number analyzed (Participants) | 1 | 0 | 0 | 1 | 2 | 5
  Change at Day 489 | -14.38 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. |  |  | -1.05 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | -1.80 (0.870) | -16.47 (28.357)
  Change at Day 534: number analyzed (Participants) | 1 | 0 | 0 | 1 | 1 | 5
  Change at Day 534 | -6.82 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. |  |  | -0.86 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | -2.34 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | -16.25 (28.463)
  Change at Day 579: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 5
  Change at Day 579 | -13.88 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. |  |  |  |  | -15.81 (28.620)
  Change at Day 624: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3
  Change at Day 624 |  |  |  |  |  | -23.45 (37.575)
  Change at Early Discontinuation: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Change at Early Discontinuation |  |  |  |  |  | 2.30 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.

14. Other Pre Specified Outcome: Change From Baseline in Log CRP Concentrations at Day 7, 14, 28, 35, 42, 56, 63, 70, 84, 129, 174, 219, 264, 309, 354, 399, 444, 489, 534, 579, 624
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Day 7, 14, 28, 35, 42, 56, 63, 70, 84, 129, 174, 219, 264, 309, 354, 399, 444, 489, 534, 579, 624
Population: Data for this outcome measure was not assessed since this measure was analyzed as per sponsor discretion as the change from baseline in CRP in this study was well demonstrated with the raw CRP data. Therefore, log transformation of CRP was not performed.
Arm/Group | Placebo | PF-04236921 1 mg | PF-04236921 10 mg | PF-04236921 30 mg | PF-04236921 100 mg | PF-04236921 250 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

15. Other Pre Specified Outcome: Change From Baseline in Absolute Neutrophil Counts at Day 7, 14, 28, 35, 42, 56, 63, 70, 84, 129, 174, 219, 264, 309, 354, 399, 444, 489, 534, 579, 624 and Early Discontinuation
Time Frame: as for outcome 13
Population: Pharmacodynamic analysis set included all enrolled participants who received at least 1 dose of study medication and had at least 1 pharmacodynamic parameter.Data collected at Early Discontinuation included those subjects who left the study early. 'N' (number of participants analyzed) = participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: 10^3 cells/millimeter (mm)^3
Arm/Group | Placebo | PF-04236921 1 mg | PF-04236921 10 mg | PF-04236921 30 mg | PF-04236921 100 mg | PF-04236921 250 mg
Number analyzed (Participants) | 8 | 5 | 6 | 6 | 5 | 7
10^3 cells/millimeter (mm)^3
  Baseline | 3.41 (1.458) | 4.13 (1.161) | 4.35 (1.203) | 4.38 (1.791) | 4.26 (1.058) | 3.13 (0.950)
  Change at Day 7 | 0.27 (0.932) | -0.16 (1.707) | -1.61 (0.936) | -0.61 (0.756) | -1.87 (0.550) | -1.08 (0.671)
  Change at Day 14 | 0.34 (0.919) | -0.71 (1.145) | -1.34 (0.586) | -0.70 (0.899) | -1.91 (0.660) | -0.78 (0.588)
  Change at Day 28: number analyzed (Participants) | 8 | 5 | 5 | 6 | 5 | 7
  Change at Day 28 | 0.24 (0.632) | -0.58 (1.828) | -0.56 (1.278) | -0.66 (0.764) | -1.91 (0.460) | -0.60 (0.637)
  Change at Day 35: number analyzed (Participants) | 8 | 5 | 5 | 6 | 5 | 7
  Change at Day 35 | 0.34 (0.987) | -0.39 (1.394) | -1.92 (1.051) | -1.28 (0.574) | -2.08 (0.756) | -0.70 (0.859)
  Change at Day 42: number analyzed (Participants) | 8 | 5 | 5 | 6 | 5 | 7
  Change at Day 42 | 0.48 (0.842) | -0.67 (1.834) | -1.19 (0.763) | -0.54 (1.094) | -1.78 (0.954) | -0.83 (0.617)
  Change at Day 56: number analyzed (Participants) | 8 | 5 | 5 | 5 | 4 | 7
  Change at Day 56 | 0.49 (1.085) | -0.79 (1.071) | -1.75 (1.024) | -1.11 (0.682) | -1.47 (0.778) | -1.27 (0.674)
  Change at Day 63: number analyzed (Participants) | 8 | 5 | 5 | 6 | 5 | 7
  Change at Day 63 | -0.45 (1.683) | -1.17 (1.742) | -1.36 (0.548) | -1.23 (0.872) | -1.69 (0.979) | -1.04 (0.657)
  Change at Day 70: number analyzed (Participants) | 8 | 5 | 5 | 5 | 5 | 7
  Change at Day 70 | 0.57 (0.883) | -1.18 (1.054) | -1.80 (0.952) | -0.48 (0.746) | -2.20 (1.218) | -1.11 (0.871)
  Change at Day 84: number analyzed (Participants) | 7 | 5 | 5 | 6 | 5 | 7
  Change at Day 84 | -0.05 (0.427) | -0.87 (1.257) | -1.77 (1.138) | -0.33 (1.740) | -1.02 (1.858) | -1.24 (0.719)
  Change at Day 129: number analyzed (Participants) | 7 | 4 | 4 | 5 | 5 | 7
  Change at Day 129 | 1.56 (2.271) | -0.35 (0.289) | -1.40 (1.424) | -0.84 (1.005) | -1.62 (0.757) | -0.60 (0.458)
  Change at Day 174: number analyzed (Participants) | 6 | 2 | 5 | 6 | 5 | 7
  Change at Day 174 | 0.49 (1.222) | -0.51 (1.944) | -1.27 (1.468) | -0.09 (2.183) | -1.25 (1.254) | -0.58 (0.254)
  Change at Day 219: number analyzed (Participants) | 6 | 2 | 5 | 6 | 5 | 6
  Change at Day 219 | 0.69 (1.071) | -0.99 (0.994) | -1.11 (1.111) | -0.75 (0.876) | -1.71 (0.906) | -0.82 (0.667)
  Change at Day 264: number analyzed (Participants) | 5 | 1 | 3 | 5 | 5 | 5
  Change at Day 264 | 0.69 (0.653) | -1.48 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | -0.87 (0.969) | -1.28 (0.857) | -1.36 (1.237) | -0.64 (0.683)
  Change at Day 309: number analyzed (Participants) | 2 | 0 | 2 | 5 | 5 | 3
  Change at Day 309 | 0.05 (0.452) |  | -2.61 (0.709) | -1.34 (0.726) | -1.01 (0.990) | -0.42 (0.726)
  Change at Day 354: number analyzed (Participants) | 2 | 0 | 1 | 5 | 5 | 5
  Change at Day 354 | 1.46 (0.296) |  | -2.02 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | -0.88 (0.448) | -1.33 (0.624) | -0.16 (0.717)
  Change at Day 399: number analyzed (Participants) | 2 | 0 | 0 | 3 | 5 | 5
  Change at Day 399 | 0.44 (0.922) |  |  | -0.61 (0.781) | 0.34 (2.056) | -0.11 (0.901)
  Change at Day 444: number analyzed (Participants) | 1 | 0 | 0 | 1 | 2 | 5
  Change at Day 444 | 0.47 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. |  |  | -0.32 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | -0.96 (2.067) | 0.11 (1.064)
  Change at Day 489: number analyzed (Participants) | 1 | 0 | 0 | 0 | 2 | 5
  Change at Day 489 | 0.68 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. |  |  |  | -1.24 (0.564) | 0.05 (0.769)
  Change at Day 534: number analyzed (Participants) | 1 | 0 | 0 | 1 | 1 | 5
  Change at Day 534 | -0.10 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. |  |  | -0.61 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | -1.07 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | -0.22 (0.685)
  Change at Day 579: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 5
  Change at Day 579 | 0.16 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. |  |  |  |  | 0.41 (0.566)
  Change at Day 624: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3
  Change at Day 624 |  |  |  |  |  | 0.10 (0.792)
  Change at Early Discontinuation: number analyzed (Participants) | 8 | 5 | 6 | 4 | 5 | 6
  Change at Early Discontinuation | 0.00 (0.498) | 0.93 (1.106) | -1.00 (0.899) | -0.69 (1.087) | -0.63 (0.849) | -0.07 (0.948)

16. Other Pre Specified Outcome: Change From Baseline in Free Interleukin-6 (IL-6) Concentrations at Day 28, 56, 84, 129, 174, 219, 264, 309, 354, 399, 444, 489, 534, 579 and 624
Description: Serum samples were analyzed for IL-6 concentrations using a validated analytical colorimetric Enzyme-Linked Immunosorbent Assay (ELISA) method.
Time Frame: Baseline, Day 28, 56, 84, 129, 174, 219, 264, 309, 354, 399, 444, 489, 534, 579, 624
Population: Pharmacodynamic analysis set included all enrolled participants who received at least 1 dose of study medication and had at least 1 pharmacodynamic parameter. n=participants evaluable for this measure at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Placebo | PF-04236921 1 mg | PF-04236921 10 mg | PF-04236921 30 mg | PF-04236921 100 mg | PF-04236921 250 mg
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 6 | 7
picogram per milliliter (pg/mL)
  Baseline | 12.55 (14.593) | 9.11 (7.204) | 17.82 (12.433) | 3.96 (3.272) | 11.75 (9.797) | 9.49 (11.744)
  Change at Day 28: number analyzed (Participants) | 9 | 6 | 5 | 6 | 6 | 7
  Change at Day 28 | 0.45 (5.383) | -2.16 (5.767) | -13.12 (13.086) | -2.40 (3.272) | -9.70 (9.147) | -7.25 (10.337)
  Change at Day 56: number analyzed (Participants) | 9 | 6 | 5 | 6 | 6 | 7
  Change at Day 56 | -2.00 (8.081) | -3.04 (6.583) | -16.14 (12.643) | -1.80 (3.342) | -10.19 (9.797) | -7.93 (11.744)
  Change at Day 84: number analyzed (Participants) | 9 | 4 | 5 | 6 | 6 | 7
  Change at Day 84 | -0.04 (14.524) | -5.60 (7.278) | -14.96 (14.406) | -2.08 (3.623) | -10.19 (9.797) | -7.29 (11.313)
  Change at Day 129: number analyzed (Participants) | 8 | 4 | 5 | 6 | 6 | 7
  Change at Day 129 | -1.25 (8.691) | -1.90 (9.291) | -13.39 (13.627) | -1.89 (3.907) | -10.19 (9.797) | -7.16 (11.507)
  Change at Day 174: number analyzed (Participants) | 7 | 2 | 5 | 6 | 6 | 7
  Change at Day 174 | 4.53 (20.905) | -4.70 (14.863) | -11.63 (12.903) | -1.34 (4.056) | -10.19 (9.797) | -7.22 (11.332)
  Change at Day 219: number analyzed (Participants) | 7 | 2 | 5 | 6 | 6 | 6
  Change at Day 219 | 4.51 (19.163) | -2.51 (16.794) | -14.23 (13.524) | -0.77 (3.830) | -10.19 (9.797) | -3.89 (7.796)
  Change at Day 264: number analyzed (Participants) | 6 | 1 | 3 | 5 | 6 | 5
  Change at Day 264 | -2.33 (14.034) | -17.94 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | -1.03 (17.395) | -1.39 (2.609) | -9.93 (9.856) | -1.33 (1.905)
  Change at Day 309: number analyzed (Participants) | 3 | 0 | 2 | 5 | 6 | 5
  Change at Day 309 | -1.36 (2.356) |  | -9.19 (18.993) | -1.67 (2.506) | -8.87 (10.655) | -1.33 (1.905)
  Change at Day 354: number analyzed (Participants) | 3 | 0 | 1 | 5 | 6 | 5
  Change at Day 354 | -1.36 (2.356) |  | -20.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | -2.34 (3.487) | -8.61 (10.701) | -1.33 (1.905)
  Change at Day 399: number analyzed (Participants) | 3 | 0 | 0 | 3 | 6 | 5
  Change at Day 399 | -1.36 (2.356) |  |  | 2.15 (4.508) | -3.74 (17.157) | -1.33 (1.905)
  Change at Day 444: number analyzed (Participants) | 1 | 0 | 0 | 1 | 3 | 5
  Change at Day 444 | -4.08 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. |  |  | 4.69 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | -8.19 (12.557) | -0.78 (1.865)
  Change at Day 489: number analyzed (Participants) | 1 | 0 | 0 | 1 | 2 | 5
  Change at Day 489 | -4.08 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. |  |  | -2.51 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | -6.31 (19.778) | -0.44 (2.157)
  Change at Day 534: number analyzed (Participants) | 1 | 0 | 0 | 1 | 1 | 5
  Change at Day 534 | -4.08 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. |  |  | -2.51 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | -20.93 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | -1.33 (1.905)
  Change at Day 579: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 5
  Change at Day 579 | -4.08 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. |  |  |  |  | -1.33 (1.905)
  Change at Day 624: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3
  Change at Day 624 |  |  |  |  |  | -0.85 (1.472)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | PF-04236921 1 mg | PF-04236921 10 mg | PF-04236921 30 mg | PF-04236921 100 mg | PF-04236921 250 mg
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/6 | 2/6 | 1/6 | 0/7
Other Adverse Events (participants affected / at risk) | 9/9 | 4/6 | 4/6 | 6/6 | 6/6 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=9) | PF-04236921 1 mg (N=6) | PF-04236921 10 mg (N=6) | PF-04236921 30 mg (N=6) | PF-04236921 100 mg (N=6) | PF-04236921 250 mg (N=7)
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=9) | PF-04236921 1 mg (N=6) | PF-04236921 10 mg (N=6) | PF-04236921 30 mg (N=6) | PF-04236921 100 mg (N=6) | PF-04236921 250 mg (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Feeling cold (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 0 | 2 | 2 | 2
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 2 | 1 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 1
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Urine analysis abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 2 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 3 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.